CLINICAL TRIAL: NCT03146572
Title: Utilizing the Primary Care Setting to Deliver a Brief Program to Enhance Parenting Behaviors
Brief Title: Primary Care and Parenting
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Society of Developmental and Behavioral Pediatrics (Unknown)
Responsible Party: Principal Investigator, Reshma Shah, MD, Assistant Professor of Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-0337_2; SDBP (Other: Society of Developmental and Behavioral Pediatrics)
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Parenting; Knowledge, Attitudes, Practice; Development, Child
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parent of child to receive intervention, Sit Down and Play
  Interventions: Behavioral: Sit Down and Play
- Control (Active Comparator): Parent will receive handout to promote positive behavior
  Interventions: Other: Handout

INTERVENTIONS:
Behavioral: Sit Down and Play — Sit Down and Play (SDP) is designed to be a brief, low-cost intervention that incorporates key theoretical constructs to elicit positive parenting behaviors. It is intended to be delivered by existing clinical staff, nonprofessionals, or volunteers during each of the eight well-child visits between 2-24 months of age while a family waits to be seen by their pediatrician in the examination room
  Other Names: Handout
  Arms: Intervention
Other: Handout — Handout providing written descriptions of strategies to encourage positive parenting behaviors
  Arms: Control

SUMMARY:
The objective of this study to evaluate potential impact of a brief, low-cost primary care-based intervention of parenting self-efficacy, knowledge, and behavior.

DETAILED DESCRIPTION:
Enriching parenting behaviors in early childhood promotes child development and offers a promising strategy to reduce future educational disparities. However, current interventions are limited by cost and have not been widely disseminated. Recognized as a target for research to improve early childhood development and subsequent school readiness skills among at-risk families, the primary care setting offers an ideal opportunity to reach the millions of children living in poverty. However, what remains unknown is how to more efficiently leverage the primary care setting to deliver a sustainable and effective preventive program to promote positive parenting behaviors and encourage early childhood development in low-income families. Therefore, the investigators designed Sit Down and Play (SDP) a brief parent-directed program delivered in the primary care setting. Modeled after the widely disseminated literacy program Reach Out and Read and grounded in social cognitive theory, SDP is intended to take place during each pediatric well-child visit occurring in a child's first two years with the goal of promoting positive parenting behaviors.

ELIGIBILITY:
Inclusion Criteria:

Parent is 18 years or older Child is present for a 6, 9, or 12 month well-child visit who attends University of Illinois at Chicago (UIC) for well-child care Adult present with child at appointment is parent/caregiver of child

Exclusion Criteria:

Parent is non-English speaking Child is acutely sick

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-02-11 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Change in Parental Knowledge | Enrollment and 7 months post-enrollment
  Change in parental knowledge regarding importance of talking with children
Change in participation in cognitively stimulating activities | Enrollment and 7 months post-enrollment
  Change in participation in cognitively stimulating activities such as reading and play as measured by the StimQ
Change in parenting self-efficacy | Enrollment and 7 months post-enrollment
  Change in perceived self-efficacy in parenting activity as measured by The Tool to Measure Parenting Self Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Shah, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States